CLINICAL TRIAL: NCT02227108
Title: A Phase 2, Multicenter, Single-arm Study of Moxetumomab Pasudotox in Pediatric Subjects With Relapsed or Refractory Pediatric Acute Lymphoblastic Leukemia (pALL) or Lymphoblastic Lymphoma of B-cell Origin
Brief Title: Study in Pediatrics With Relapsed or Refractory Pediatric Acute Lymphoblastic Leukemia (pALL) or Lymphoblastic Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated prior to a planned interim analysis based on lack of required efficacy in the first 32 participants enrolled.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-CAT-8015-1036
Record Dates: First submitted 2014-08-21; First posted 2014-08-27 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: B-Cell Pediatric ALL
Keywords: pediatric cancer,pediatric acute lymphoblastic leukemia, lymphoblastic lymphoma, B-cell leukemia, ALL, moxetumomab pasudotox, CD22
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, B-Cell | interventions — immunotoxin HA22

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Moxetumomab Pasudotox 40 mcg/kg (Experimental): Participants received 6 doses of moxetumomab pasudotox 40 microgram per kilogram (mcg/kg) intravenous infusion over 30 minutes every other day (Days 1, 3, 5, 7, 9, and 11) in 21-day treatment cycles until completion of a maximum of 6 cycles of therapy.
  Interventions: Drug: Moxetumomab Pasudotox

INTERVENTIONS:
Drug: Moxetumomab Pasudotox — Participants received 6 doses of moxetumomab pasudotox 40 microgram per kilogram (mcg/kg) intravenous infusion over 30 minutes every other day (Days 1, 3, 5, 7, 9, and 11) in 21-day treatment cycles until completion of a maximum of 6 cycles of therapy.
  Other Names: CAT-8015

SUMMARY:
The primary objective of this study is to evaluate the efficacy of moxetumomab pasudotox in pediatric participants with relapsed or refractory B-cell acute lymphoblastic leukemia (ALL) or B-cell lymphoblastic lymphoma.

DETAILED DESCRIPTION:
This is a global, multicenter, open-label, single-arm Phase 2 study to evaluate the efficacy and safety of moxetumomab pasudotox monotherapy in pediatric participants with relapsed or refractory B-cell ALL or B-cell lymphoblastic lymphoma. Participants will be enrolled at sites in North America, Europe, and Australia. This is an approximate 35 month study.

ELIGIBILITY:
Inclusion Criteria -

1. Between the ages of greater or equal to (≥) 6 months and less than (<) 18 years of age
2. Must have histologically proven B-cell acute lymphoblastic leukemia (ALL) or B-cell lymphoblastic lymphoma with marrow involvement
3. All participants (both ALL and participants with lymphoblastic lymphoma) must have M2 or M3 bone marrow classification
4. Disease status: a) Participants must have relapsed or refractory disease b) In the event of relapse after prior allogeneic hematopoietic stem cell transplant (HSCT), participants must be at least 3 months post-transplant and have no evidence of active graft-vs-host disease, and must have been off immunosuppression for at least 4 weeks, c) Must have resolution of the acute toxic effects to less than or equal to (≤) Grade 2 from prior chemotherapy before entry, in the opinion of the investigator
5. Participants with the following central nervous system (CNS) 1 or 2 status are eligible only in the absence of neurologic symptoms
6. Female participants of childbearing potential and post-pubertal male participants must use an approved method of contraception for the study.

Exclusion Criteria

1. Concurrent enrollment in another clinical study for cancer treatment, unless the subject is in the follow-up period from a previous study.
2. Isolated testicular or CNS ALL
3. Participants with mixed-lineage leukemia (MLL) gene rearrangement
4. Inadequate Hepatic function
5. Inadequate Renal function
6. Radiologically-detected CNS lymphoma
7. Participants with clear laboratory or clinical evidence of disseminated intravascular coagulation (DIC)
8. Hyperleukocytosis or rapidly progressive disease that would compromise ability to complete study therapy
9. QT interval corrected using Fridericia's formula (QTcF) greater than or equal to a Grade 2, confirmed by 2 additional seperate electrocardiographs (ECG's) within 28 days prior to starting study drug. The initial screening ECG need not be repeated for confirmation if the QTcF interval is <481 milliseconds.
10. Pregnant or breast-feeding females
11. Prior treatment with CAT-3888 (BL22), moxetumomab pasudotox, or any pseudomonas-exotoxin-containing compound
12. Prior treatment with any anticancer biologic therapy within 2 weeks prior to starting study drug, including but not limited to therapeutic monoclonal antibodies or antibody-drug conjugates
13. Systemic chemotherapy ≤ 2 weeks (6 weeks for nitrosoureas) and radiation therapy ≤ 3 weeks prior to starting study drug
14. Clinically significant ophthalmologic findings (evidence of retinal damage or injury) during the screening
15. Presence of a second invasive malignancy
16. Uncontrolled pulmonary infection, presence of pulmonary edema
17. Serum albumin < 2 gram per deciliter (g/dL). Albumin infusions for correction of hypoalbuminemia are allowed, but cannot have administered within 7 days prior to start of study drug
18. Radioimmunotherapy within 2 years prior to study start of study drug
19. Participants with prior history of thrombotic microangiopathy or hemolytic uremic syndrome (HUS)
20. T-cell ALL or T-cell lymphoblastic lymphoma
21. Participants currently receiving high-dose estrogen therapy defined as >0.625 milligram per day (mg/day) of an estrogen compound or within 2 weeks prior to starting study drug.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune Inc. Medimmune Inc., Study Director — MedImmune LLC
Locations (21):
- United States (10):
  - Research Site, Phoenix, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Chicago, Illinois
  - Research Site, Bethesda, Maryland
  - Research Site, Kansas City, Missouri
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Parkville
  - Research Site, Westmead
- Research Site, Edmonton, Alberta, Canada
- France (3):
  - Research Site, Lyon
  - Research Site, Paris
  - Research Site, Vandœuvre-lès-Nancy
- Research Site, Rome, Italy
- Research Site, Rotterdam, Netherlands
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid
- Research Site, Bristol, United Kingdom

REFERENCES:
- [Background] Mussai F, Campana D, Bhojwani D, Stetler-Stevenson M, Steinberg SM, Wayne AS, Pastan I. Cytotoxicity of the anti-CD22 immunotoxin HA22 (CAT-8015) against paediatric acute lymphoblastic leukaemia. Br J Haematol. 2010 Aug;150(3):352-8. doi: 10.1111/j.1365-2141.2010.08251.x. Epub 2010 Jun 7. PMID 20528877

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were screened, of which 5 did not meet eligibility criteria and were considered as screen failures; the remaining 32 participants entered into the study and 30 participants were treated with moxetumomab pasudotox.
Groups:
- Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg): Participants received 6 doses of moxetumomab pasudotox 40 mcg/kg intravenous infusion over 30 minutes every other day (Days 1, 3, 5, 7, 9, and 11) in 21-day treatment cycles until completion of a maximum of 6 cycles of therapy.
Period: Overall Study
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Started | 32
Treated | 30
Completed | 1
Not Completed | 31
Not completed — Did not receive treatment | 2
Not completed — Other | 3
Not completed — Progressive disease | 17
Not completed — Initiation of alternative therapy | 2
Not completed — Investigator discretion | 1
Not completed — Adverse Event | 6

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who entered the study.
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.5 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Complete Response (CRc)
Description: The CRc is defined as achieving complete response (CR), or CR with incomplete count recovery [CRi]) in participants with relapsed or refractory B-cell ALL or B-cell lymphoblastic lymphoma. Complete response (CR) as per International Working Group (IWG) is complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Morphologic CR with incomplete blood count recovery (CRi) is defined as the above CR criteria without specified blood counts. The efficacy assessments were evaluated as per investigator assessment.
Time Frame: Prior to Cycle 1, and prior to every cycle, at the end of treatment, at post-treatment follow-up visits, and at the end of the study, up to 1 year
Population: Efficacy evaluable population included all participants who received any amount of moxetumomab pasudotox and completed a baseline disease assessment and had at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
percentage of participants | 10.7 [2.3 to 28.2]

2. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD)-Negative CRc Rate
Description: The MRD-negative CRc rate was defined as the percentage of participants who achieved CRc and became MRD-negative as determined by flow cytometry performed by a central analysis laboratory. The CRc is defined as complete response (CR), or complete response with incomplete count recovery (CRi). Complete response (CR) as per International Working Group (IWG) is complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Morphologic CR with incomplete blood count recovery (CRi) is defined as the above CR criteria without specified blood counts.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
percentage of participants | 0

3. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR, defined as the percentage of participants with CRc or partial response (PR), was estimated; the Clopper Pearson (Exact) 95% CI was calculated. The CRc is defined as complete response (CR), or complete response with incomplete count recovery (CRi). Complete response (CR) as per International Working Group (IWG) is complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Morphologic CR with incomplete blood count recovery (CRi) is defined as the above CR criteria without specified blood counts.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
percentage of participants | 28.6 [13.2 to 48.7]

4. Secondary Outcome: Time to Overall Response
Description: Time to overall response was evaluated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
months | 0.66 [0.53 to 0.76]

5. Secondary Outcome: Best Overall Response (BOR)
Description: The best overall response was calculated, based upon the disease assessments recorded during the study visits, and summarized with the number and percentage of participants for the following categories: CRc, PR, HA, SD, PD, and not evaluable. Overall best response is the best response observed for a participant during the study based on International Working Group (IWG) Response Criteria for malignant lymphoma. Complete response (CR) as per IWG is complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. PR is a minimum of 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses and no increase in the size of other nodes and in size of liver or spleen. Stable disease (SD) is when a participant fails to attain the criteria needed for a CR or PR, but does not fulfill those for PD.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
percentage of participants
  Composite complete response | 10.7
  Partial response | 17.9
  Hematological activity | 7.1
  Stable disease | 21.4
  Progressive disease | 39.3
  No evaluation available | 3.6

6. Secondary Outcome: Bone Marrow Blast Percentage Change
Description: Change in bone marrow blast percentage from baseline was evaluated. If the percentage (%) blasts (at least 200 cells counted) is less than (<) 5%, it is considered as M1, 5 to 25% considered as M2, greater than (>) 25% considered as M3. Stages with the higher blasts relate to worse outcomes.
Time Frame: as for outcome 1
Population: The intent to treat (ITT) population included all participants who entered the study. Here, number of participants analysed, "N" included evaluable participants for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 26
percentage of participants
  Baseline M1, post-baseline M1 | 0
  Baseline M1, post-baseline M2 | 0
  Baseline M1, post-baseline M3 | 3.8
  Baseline M2, post-baseline M1 | 0
  Baseline M2, post-baseline M2 | 0
  Baseline M2, post-baseline M3 | 7.7
  Baseline M3 post-baseline M1 | 3.8
  Baseline M3 post-baseline M2 | 11.5
  Baseline M3 post-baseline M3 | 73.1

7. Secondary Outcome: Percentage of Participants Who Became Eligible to Receive an Stem Cell Transplant (SCT) After Treatment With Moxetumomab Pasudotox
Description: The percentage of participants who became eligible for SCT after treatment with moxetumomab pasudotox were provided. The Clopper Pearson (Exact) 95% CI was calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
percentage of participants | 0

8. Secondary Outcome: Time to Transplant to Receive an Stem Cell Transplant (SCT) After Treatment With Moxetumomab Pasudotox
Description: The time to SCT was defined as the duration from the start of treatment with moxetumomab pasudotox until the date when the subject became eligible for SCT. The time to SCT was to be summarized using the Kaplan-Meier method, and was only to be evaluated for the subgroup of subjects who became eligible for SCT after treatment with moxetumomab pasudotox.
Time Frame: as for outcome 1
Population: Efficacy population included participants who received moxetumomab pasudotox, completed a baseline disease assessment and had at least one post-baseline assessment. Since study was terminated prematurely, no participant received SCT after treatment with moxetumomab pasudotox, hence data were not collected for this Outcome measure.
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 0

9. Secondary Outcome: Percentage of Participants Who Were Neutropenic at Study Entry and Who Experienced Hematologic Activity (HA)
Description: The percentage of participants who were neutropenic at study entry and experienced HA after treatment with moxetumomab pasudotox was evaluated. The Clopper Pearson (Exact) 95% CI was calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
percentage of participants | 3.6

10. Secondary Outcome: Duration of Complete Response (DOCR)
Description: DOCR was defined as the duration from the first documentation of CRc to the first documented disease progression.The CRc is defined as achieving complete response (CR), or CR with incomplete count recovery [CRi]) in participants with relapsed or refractory B-cell ALL or B-cell lymphoblastic lymphoma. Kaplan-Meier method was used for evaluation.
Time Frame: as for outcome 1
Population: Efficacy evaluable population included all participants who received any amount of moxetumomab pasudotox and completed a baseline disease assessment and had at least one post-baseline disease assessment. Here, number of participants analysed, "N" included evaluable participants for this outcome measure.
Measure: Number; unit: months
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 1
months | 1.97 [0 to 0]

11. Secondary Outcome: Duration of Overall Response (DOR)
Description: DOR was to be defined as the duration from the first documentation of overall response to the first documented disease progression. Kaplan-Meier method was used for evaluation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
months | 0.95 [0.59 to 1.97]

12. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was measured from the start of treatment with moxetumomab pasudotox until the first documentation of disease progression or death due to any cause, whichever occurred first. Kaplan-Meier method was used for evaluation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
months | 1.4 [0.3 to 8.4]

13. Secondary Outcome: Overall Survival (OS)
Description: OS was determined as the time from the start of treatment with moxetumomab pasudotox until death due to any cause. For participants who were alive at the end of the study or lost to follow-up, OS was censored on the last date when the participant was known be alive. Kaplan-Meier method was used for evaluation.
Time Frame: Baseline to end of study or last contact date, up to 1 year
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 28
months | 3.6 [0.4 to 9.8]

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: Treatment-emergent adverse events (TEAEs), were defined as events present at baseline that worsened in intensity after administration of investigational product or events absent at baseline that emerged after administration of study drug.
Time Frame: Baseline up to 30 days after the last dose of study drug, up to 1 year
Population: Safety population includes all participants who received any amount of moxetumomab pasudotox.
Measure: Number; unit: participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 30
participants
  TEAEs | 30
  TESAEs | 16

15. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as Treatment-Emergent Adverse Events (TEAE)
Description: Laboratory tests were grouped according to hematology, serum chemistry, and urinalysis. Laboratory abnormalities with toxicity grades according to NCI CTCAE Version 4.03 were derived according to laboratory values and reported as treatment-emergent adverse events.
Time Frame: Baseline up to 30 days after the last dose of study drug, up to 1 year
Population: Safety population includes all participants who received any amount of moxetumomab pasudotox.
Measure: Number; unit: participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 30
participants
  Anaemia | 11
  Febrile neutropenia | 7
  Haemolytic uraemic syndrome | 4
  Thrombocytopenia | 1
  Platelet count decreased | 9
  Neutrophil count decreased | 6
  White blood cell count decreased | 5
  Lymphocyte count decreased | 2
  International normalised ratio increased | 1
  Alanine aminotransferase increased | 11
  Aspartate aminotransferase increased | 8
  Gamma-glutamyltransferase increased | 4
  Blood bilirubin increased | 2
  Blood creatinine increased | 2
  Blood lactate dehydrogenase increased | 2
  Bilirubin conjugated | 1
  Blood albumin decreased | 1
  Blood urea increased | 1
  Glucose tolerance increased | 1
  Hypoalbuminaemia | 6
  Hypocalcaemia | 6
  Hypokalaemia | 5
  Hyponatraemia | 5
  Hyperglycaemia | 4
  Hypophosphataemia | 3
  Hypermagnesaemia | 1
  Hypomagnesaemia | 1
  Hepatic function abnormal | 1
  Proteinuria | 1

16. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Participants were evaluated for ECG abnormalities.
Time Frame: Baseline up to 30 days after the last dose of study drug, up to 1 year
Population: Safety population includes all participants who received any amount of moxetumomab pasudotox.
Measure: Number; unit: participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 30
participants | 0

17. Secondary Outcome: Number of Participants With Abnormal Vital Signs Reported as Treatment-Emergent Adverse Events (TEAEs)
Description: Participants who experienced vital signs abnormalities recorded as TEAEs were reported.
Time Frame: Baseline up to 30 days after the last dose of study drug, up to 1 year
Population: Safety population includes all participants who received any amount of moxetumomab pasudotox.
Measure: Number; unit: participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 30
participants
  Pyrexia | 16
  Dyspnoea | 6
  Hypoxia | 4
  Hypertension | 8
  Hypotension | 4
  Weight decreased | 1
  Weight increased | 10
  Bradycardia | 7
  Sinus bradycardia | 1
  Sinus tachycardia | 3
  Tachycardia | 3

18. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) and Neutralizing Antibodies (NAb)
Description: Immunogenicity assessment included determination of antidrug (moxetumomab pasudotox) antibodies and neutralizing antidrug antibodies in serum samples. Titers and specificity were determined for NAb-positive participants. Specificity were observed in participants who had ADAs directed to the PE38 domain of moxetumomab pasudotox and increase in titers were observed in participants who tested ADA-positive at baseline. Moxetumomab pasudotox ADA-titer is a validated immunoassay, which determines titers or levels of ADAs present in ADA-positive samples.
Time Frame: Prior to the Start of Each Cycle for Cycles 1, 2, 3, and Subsequent Odd-Numbered Cycles, End of Treatment, and 30 Day Follow-up Visit, up to 1 year
Population: Safety population includes all participants who received any amount of moxetumomab pasudotox. Here, number of participants analysed, "N" included participants with at least one post-baseline sample.
Measure: Number; unit: participants
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 23
participants
  Anti-drug Antibody (ADA) | 13
  Neutralizing Antibodies (NAb) | 13
  Increase in Titers | 3
  Specificity | 13

19. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to Infinity (AUC0-inf) After the First Dose of Cycle 1
Description: AUC (0-infinity) = Area under the serum concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (tinfinity). It was calculated by extrapolating the concentrationtime curve from time zero to infinity using the linear/log trapezoidal rule.
Time Frame: Pre-infusion, end of infusion (EOI); 1, 3, and 6 hours post-infusion of Day 1 of Cycle 1
Population: Safety population who provided at least one measurable Pharmacokinetic concentration. Here, number of participants analysed, "N" included evaluable participants for this outcome measure.
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7
hour*nanogram per milliliter (hr*ng/mL) | 1200 (224)

20. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to Last Quantifiable Concentration [AUC0-last] After the First Dose of Cycle 1
Description: AUC is a measure of systemic drug exposure, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample. AUC0-t is defined as AUC from time zero to the last data point above the lower limit of quantification.
Time Frame: Pre-infusion, end of infusion (EOI); 1, 3, and 6 hours post-infusion at Day 1 of Cycle 1
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 21
hour*nanogram per milliliter (hr*ng/mL) | 794 (239)

21. Secondary Outcome: Maximum Observed Drug Concentration in Plasma (Cmax) After the First Dose of Cycle 1
Description: Cmax refers to the highest measured drug concentration which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Time Frame: Pre-infusion, end of infusion (EOI); 1, 3, and 6 hours post-infusion at Day 1 of Cycle 1
Population: Safety population who provided at least one measurable Pharmacokinetic concentration.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 26
nanogram per milliliter | 457 (128)

22. Secondary Outcome: Time to Reach Maximum Drug Concentration in Plasma (Tmax) After the First Dose of Cycle 1
Description: Tmax refers to the time after dosing when a drug attains its highest measurable concentration (Cmax). It is obtained by collecting a series of blood samples at various times after dosing, and measuring them for drug content.
Time Frame: Pre-infusion, end of infusion (EOI); 1, 3, and 6 hours post-infusion at Day 1 of Cycle 1
Population: Safety population who provided at least one measurable Pharmacokinetic concentration.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 26
hour | 0.54 (0.05) [0.50 to 0.75]

23. Secondary Outcome: Terminal Phase Elimination Half Life (t1/2) After the First Dose of Cycle 1
Description: Terminal phase elimination half-life is the time measured for the serum/plasma concentration to decrease by one half, calculated as natural logarithmic (log)-transformed (ln) value of 2 divided by elimination rate constant (lambda); that is [ln(2)/lambda]. Elimination rate constant (lambda) was estimated via linear regression of the time versus log concentration.
Time Frame: Pre-infusion, end of infusion (EOI); 1, 3, and 6 hours post-infusion at Day 1 of Cycle 1
Population: as for outcome 19
Measure: Median (Full Range); unit: hour
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7
hour | 1.02 (0.213) [0.820 to 1.44]

24. Secondary Outcome: Systemic Clearance (CL) After the First Dose of Cycle 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. The total systemic clearance after intravenous dose was estimated by dividing the total administered dose by the plasma Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]).
Time Frame: Pre-infusion, end of infusion (EOI); 1, 3, and 6 hours post-infusion at Day 1 of Cycle 1
Population: as for outcome 19
Measure: Mean (Full Range); unit: milliliter per hour per kilogram
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Number analyzed (Participants) | 7
milliliter per hour per kilogram | 34.4 (5.72) [24.4 to 41.8]

ADVERSE EVENTS:
Time Frame: The period immediately following the time that written informed consent is obtained through Day 30 after the last dose
Arm/Group | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg)
Serious Adverse Events (participants affected / at risk) | 16/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg) (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 4 (4)
Vision blurred (Eye disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Device related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxetumomab Pasudotox 40 Microgram Per Kilogram (mcg/kg) (N=30)
Anaemia (Blood and lymphatic system disorders) | 11 (29)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (13)
Sinus tachycardia (Cardiac disorders) | 3 (6)
Tachycardia (Cardiac disorders) | 3 (3)
Periorbital oedema (Eye disorders) | 3 (3)
Vision blurred (Eye disorders) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 3 (5)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (10)
Vomiting (Gastrointestinal disorders) | 4 (4)
Face oedema (General disorders) | 4 (5)
Fatigue (General disorders) | 2 (3)
Oedema peripheral (General disorders) | 5 (8)
Pyrexia (General disorders) | 12 (40)
Pneumonia (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 11 (45)
Aspartate aminotransferase increased (Investigations) | 8 (34)
Blood bilirubin increased (Investigations) | 2 (4)
Blood creatinine increased (Investigations) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 4 (18)
Lymphocyte count decreased (Investigations) | 2 (4)
Neutrophil count decreased (Investigations) | 6 (21)
Platelet count decreased (Investigations) | 8 (59)
Weight increased (Investigations) | 10 (21)
White blood cell count decreased (Investigations) | 5 (24)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (12)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 6 (11)
Hypocalcaemia (Metabolism and nutrition disorders) | 6 (28)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (27)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (12)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 12 (22)
Paraesthesia (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 8 (12)
Hypotension (Vascular disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
The study was terminated prior to a planned interim analysis based on lack of required efficacy in the first 32 participants enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.